CLINICAL TRIAL: NCT04029103
Title: Evaluation of The Effectiveness of Mobile Diabetic Foot Personal Care System (m-DAKBAS) in Diabetic Individuals
Brief Title: Evaluation of The Effectiveness of m-DAKBAS on Foot Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanko University (Other)
Collaborators: Koç University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SankoM
Record Dates: First submitted 2019-06-26; First posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Diabetic Foot; Foot Ulcer, Diabetic; Health Knowledge, Attitudes, Practice
Keywords: Diabetic foot; health technology; mobile application
MeSH Terms: conditions — Diabetic Foot; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- used m-DAKBAS (Active Comparator): m-DAKBAS application was downloaded to the mobile phones of the participants who met the research criteria and accepted to participate in the study; the participants were given a username and a password for the confidentiality. They were instructed how to use the application after a number of trials.
  The participants were asked to send their blood sugar levels each time they measured it and foot observations daily through the application. Using the admin panel, the researcher followed the participants' frequency of using the application and the data they sent throughout 24 weeks and tried to find solutions to the problems experienced (for example: hyperglycaemia, insulin dosage adjustments). The participants were provided with feedback in line with these data; SMS reminders were sent if the tasks were not completed.
  Interventions: Other: knowledge, behaviour, self efficacy
- not used m-DAKBAS (Experimental): The participants who met the research criteria and accepted to participate in the study were given training via verbal instruction about the information in the content of m-DAKBAS (definition of Diabetic Foot, risk factors, protective precautions, daily foot care)
  Interventions: Other: knowledge, behaviour, self efficacy

INTERVENTIONS:
Other: knowledge, behaviour, self efficacy — Knowledge, behavior and self-efficacy of both groups were measured before and after the study.

SUMMARY:
Aim: To develop the Mobile Diabetic Foot Personal Care System (m-DAKBAS) related to foot care for diabetic individuals and to evaluate its effectiveness.

Method: The study involved 88 patients who applied to the Diabetes Polyclinic (intervention=44; control=44). While the intervention group used m-DAKBAS (for 6 months), the control group was provided with a verbal foot care training once, as a standardized procedure of the hospital. Data were collected using the "Socio-demographic Form", "Diabetic Foot Knowledge Form - DFKF", "Foot Self Care Behaviours Scale -FSCBS", "Diabetic Foot Care Self Efficacy Scale - DFCSES", and "m-DAKBAS Assessment Form".

DETAILED DESCRIPTION:
Diabetic foot, one of the important complications of diabetes, is a health problem that affects quality of life in a negative way, that has high treatment and care costs and mortality rates, long hospitalization duration and thus with all these aspects a psychological, physical, social and economic priority. Despite all these, diabetic foot complications and amputations could be decreased with the help of a good foot care, education and a multidisciplinary team work. Mobile technologies have been continuously increasing worldwide for the management of diabetes, and the use of these technologies is recommended by international institutions as well.

Therefore, the purpose of this study is to develop a Turkish mobile application that would increase patients' knowledge levels about foot health and care, improve their behaviours and self-efficacy, and evaluate its effectiveness so that it could be possible to prevent foot ulcer and the related amputations in individuals with diabetes. The Mobile Diabetic Foot Personal Care System (m-DAKBAS) developed for this purpose enables to increase individuals' self-confidence, improve communication with the health personnel, involve patients in their own care in an interactive way, and take responsibility.

The usability of the application was indicated by the patients' feedback, and in line with the purpose of the mobile application, improvements in the patients' knowledge, behaviours and self-efficacy about foot care in diabetes.

ELIGIBILITY:
Inclusion Criteria:

* having a diagnosis history of >1 year;
* having Type 1 or Type 2 diabetes;
* having a mobile phone with Android or IOS operating system;

Exclusion Criteria:

* having visual impairment,
* hand skill problem, difficulty in communication, or mental insufficiency;
* currently having foot ulcer.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-07-29 (Actual)

PRIMARY OUTCOMES:
Knowledge | before the intervention- Immediately after the intervention
  Diabetic Foot Knowledge Form (DFKF) included 20 questions that aim to measure the knowledge level of individuals with diabetes about diabetic foot and foot care. The questions had three options (True, False, I don't know). Each correct answer was scored 1 point. Higher scores indicate higher knowledge levels
Behaviour | before the intervention- Immediately after the intervention
  Foot Self Care Behaviours Scale is composed of 15 items which were assessed as 1=Never, 2=Rarely, 3=Sometimes, 4=Frequently, 5=Always). Scores range between 15 and 75. Higher scores indicate better self care behaviours
self-efficacy | before the intervention- Immediately after the intervention
  Diabetic Foot Care Self Efficacy Scale has nine items which are rated on an 11-item visual scale that range from 0=I find it totally insufficient and 10= I find it totally sufficient. Scores to be obtained from the scale range between 0 and 90. Higher scores indicate higher self-efficacy

CONTACTS AND LOCATIONS:
Locations (1):
- SANKO University, Şehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
the article has been sent to the journal for publication
Supporting Information: Study Protocol
Time Frame: after research published